CLINICAL TRIAL: NCT06605586
Title: A Phase 1b/2 Trial with Tasquinimod in Patients with Myelofibrosis (primary, Post-PV or PostET) Refractory to or Intolerant for JAK2 Inhibition: the TasqForce Trial
Brief Title: Tasquinimod in Patients with Myelofibrosis Refractory to or Intolerant for JAK2 Inhibition
Acronym: HOVON 172 MF
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO172; 2024-511565-11-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-01; First posted 2024-09-20 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — tasquinimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tasquinimod (Experimental): Patients will be treated with tasquinimod capsules 0.5 mg/day for 14 days (half cycle) and then capsules of 1 mg/day for the remaining 14 days in the first cycle. In consecutive 28-day cycles 1 mg/day (or if 1 mg/day is not tolerated, reduction to 0.75 or 0.5 mg/day is allowed, followed by dose re-escalation whenever possible). Patients will be treated for a maximum period of 24 weeks (6 cycles).
  Interventions: Drug: Tasquinimod

INTERVENTIONS:
Drug: Tasquinimod — treatment with tasquinimod capsules once daily

SUMMARY:
The goal of this clinical trial is to learn if therapy can be improved in patients with myelofibrosis (MF) who have primary resistance or who have progressed after treatment with a Janus kinase (JAK) inhibitor or are intolerant for this category of drugs.

The main questions it aims to answer are:

* To evaluate the feasibility and safety of once daily dose of tasquinimod for 24 weeks (6 cycles)
* To determine the optimal dose

Patients will be treated once daily with tasquinimod for a maximum period of 24 weeks (6 cycles).

During the study most (diagnostic) procedures are part of the standard of care. Different from standard of care:

* Participation may lead to extra visits to the outpatient clinic
* Additional blood will be drawn when blood is already taken per standard of care
* Bone marrow sampling at entry and at the end of the trial
* MRI scans (or CT-scans) have to be performed
* Quality-of-life questionnaires have to be filled out

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PMF or Post-PV MF or Post-ET MF based on a bone marrow (BM) biopsy not older than 6 months, according to the 2016 World Health Organization.
* Refactory or intolerant to treatment with an approved JAK inhibitor or ineligible for JAK inhibitor treatment.
* MF classified as Intermediate-1 with disease-related symptoms (e.g. symptomatic splenomegaly), Intermediate-2 or high-risk by Dynamic International Prognostic Scoring System Plus
* Spleen ≥5 cm below costal margin as measured by palpation.
* Age ≥18 years.
* Peripheral blood blast count of <10%.
* WHO/ECOG performance status of 0, 1, or 2.
* Able to swallow and retain oral medication.
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests.
* Negative pregnancy test at study entry for women of childbearing potential. Women of child-bearing potential and sexually active males must be willing and able to use highly effective methods of contraception, during treatment, and for 4 months and 6 months respectively, after study treatment.
* Patient is capable of giving informed consent.
* Written informed consent.

Exclusion Criteria:

* Patients eligible for hematopoietic stem cell transplantation (suitable candidate and a suitable donor is available).
* Splenectomy.
* Splenic irradiation within the last 6 months.
* Prior allogeneic stem cell transplantation.
* Following laboratory values within 14 days prior to registration:

  * Absolute Neutrophil Count (ANC) <0.5 x 109/L without G-CSF support
  * Platelet count <25 x 109/L without platelet transfusion
  * Serum creatinine >1.5 x Upper limit of normal (ULN) or GFR <30 ml/min
  * Serum amylase and lipase >1.5 x ULN
  * Alanine aminotransferase (ALT) ≥2.5 x ULN
  * Total bilirubin >1.5 times the upper limit of the normal range (ULN), unless elevated bilirubin is due to unconjugated hyperbilirubinemia from Gilbert's syndrome or related to MF
* Known active (acute or chronic) Hepatitis A, B, or C; and Hepatitis B and C carriers, HIV.
* Prior history of chronic liver disease (eg, chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemachromatosis).
* Patients with any other prior malignancies are not eligible, except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which subject has been disease-free for at least 5 years.
* Failure to have fully recovered (i.e. to CTCAE Grade 1 or previous baseline) from clinically significant adverse effects of prior chemotherapy (examples of adverse effects that are not clinically significant include alopecia and lymphopenia).
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of tasquinimod (e.g., ulcerative diseases, pancreatitis uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* Evidence of severe or currently uncontrolled cardiovascular condition (e.g. cardiac amyloidosis, pulmonary embolism, angina, hypertension, peripheral vascular disease, congestive heart failure class III or IV of the NYHA classification (appendix F), cardiac arrhythmia, acute coronary syndrome, myocardial infarction, cerebrovascular accident, major hemorrhage, intracranial hemorrhage, transient ischemic attack, or limb claudication) within 6 months prior to registration.
* Patients with clinically significant bacterial, fungal, parasitic or viral infection which require therapy. Patients with acute bacterial infections requiring antibiotic use should delay screening/ enrollment until the course of antibiotic therapy has been completed.
* Any chemotherapy, immunomodulatory drug therapy (eg, thalidomide, interferon-alpha), anagrelide, immunosuppressive therapy, corticosteroids >10 mg/day prednisone or equivalent, or growth factor treatment (eg, erythropoietin), or hormones (eg, androgens, danazol) within 2 weeks prior to initiation of tasquinimod; erythropoetin use within 28 days prior to initiation of tasquinimod. The only chemotherapy allowed will be hydroxyurea which has to be stopped within 1 day prior to initiation of tasquinimod.
* Treatment with fedratinib within 7 days, or momelotinib within 2 days prior to initiation of tasquinimod. For ruxolitinib no wash-out period is required before start of tasquinimod.
* Any investigational treatment for MF within 2 weeks or 5 half-lives whichever is shorter.
* History of severe hypersensitivity reaction to any component of tasquinimod.
* Systemic treatment within 14 days prior to the initiation of tasquinimod with any of the moderate or strong inhibitor, or moderate or strong inducer of cytochrome P-3A4 (CYP3A4)
* Need for ongoing therapy with drug substances of narrow therapeutic range that are metabolized mainly by CYP3A4
* Need for ongoing therapy with drug substances of narrow therapeutic range metabolized mainly by CYP1A2
* Ongoing treatment with vitamin K antagonist, unless the INR is ≤ 3.0
* Prior treatment with tasquinimod.
* Major surgery within 3 months.
* Pregnant or breast feeding (lactating) women.
* Any other condition that would, in the Investigator's judgment, contraindicate subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures e.g. any uncontrolled disease such as pulmonary disease, infection or seizure disorder; intestinal obstruction, inability to swallow medication, any altered mental status or psychiatric condition that would interfere with the understanding of the informed consent
* Current participation (during interventional treatment) in another clinical trial.
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
SVR35W24 | 24 weeks after start treatment
  Proportion of patients with at least 35% reduction in spleen volume from baseline at Week 24 (SVR35W24) as measured by magnetic resonance imaging (MRI) or computed tomography (CT) scan, per International Working Group (IWG) criteria, based on MRI review.
DLT phase I | From enrollment until 28 days after start treatment
  To determine the dose limiting toxicity (DLT) of tasquinimod. Pre-defined adverse events (AEs) that occur within 28 days of the start of study treatment will be considered a DLT, unless the AE is definitely unrelated to tasquinimod.

SECONDARY OUTCOMES:
RBC transfusions | Until end of protocol treatment after 24 weeks
  Red blood cell (RBC) transfusion (number of packed cells) during tasquinimod treatment.
Changes in variant allele frequency | Until end of protocol treatment after 24 weeks
  To determine the changes in variant allele frequency (VAF) of MPN driver genes after tasquinimod treatment by single cell and bulk DNA sequencing.
Change in splenomegaly | Until end of protocol treatment after 24 weeks
  Proportion of patients with at least 50% reduction in palpable splenomegaly from baseline per IWG criteria.
Change in spleen volume by MRI review | Until end of protocol treatment after 24 weeks
  Proportion of patients with at least 35% reduction in spleen volume from baseline (SVR35) as measured by MRI or CT scan, per IWG criteria, based on MRI review.
Changes of total symptom score | Until end of protocol treatment after 24 weeks
  Proportion of patients with at least 50% reduction in total symptom score (TSS) after 24 weeks from baseline as measured by MPN-SAF TSS.
Changes in bone marrow fibrosis | Until end of protocol treatment after 24 weeks
  Reduction in grade of bone marrow fibrosis from baseline as measured by the European consensus grading system.
Safety | until 30 days following the last dose of tasquinimod as protocol treatment
  Safety and toxicity as defined by type, frequency and severity of adverse events as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Overall survival | Until 3 years after enrollment
  Overall survival, as defined from date of registration until date of death from any cause.
Anemia response | Until end of protocol treatment after 24 weeks
  Anemia response based on transfusion dependency per IWG criteria for MF

OTHER OUTCOMES:
Plasma concentrations | Until end of protocol treatment after 24 weeks
  Plasma concentrations of tasquinimod

CONTACTS AND LOCATIONS:
Overall Officials: Peter te Boekhorst, Dr., Principal Investigator — Erasmus Medical Center
Locations (6):
- DE-Aachen-UKAACHEN, Aachen, Germany
- Netherlands (5):
  - NL-Amsterdam-AmsterdamUMC, Amsterdam
  - NL-Groningen-UMCG, Groningen
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Utrecht-UMCUTRECHT, Utrecht

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: HOVON website — http://www.hovon.org